CLINICAL TRIAL: NCT02853630
Title: A Multicentric, Randomized, Open Label Study on Comparison of Pancreatic Beta Cell Recovery and Preservation in Type 2 Diabetic Patients Treated With DPP-4 Inhibitor (Vildagliptin) and Metformin
Brief Title: A Clinical Trial to Study the Effects of Two Drugs, Vildagliptin and Metformin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237AIN04; CTRI/2014/01/004301 (Other: Clinical Trail Registry - India)
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: TYpe 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): Tablet Metformin 1000 - 2500 mg/day for 96 weeks
  Interventions: Drug: Metformin
- Vildagliptin (Experimental): Tablet Vildagliptin 100mg/day for 96 weeks
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Metformin — Participant will be instructed to take Metformin tablets as per instructions given by the physician.
  Arms: Metformin
Drug: Vildagliptin — Participant will be instructed to take one tablet of Vildagliptin 50mg per day, 30 minutes after breakfast in the morning and second tablet at night, 30 minutes after dinner
  Arms: Vildagliptin

SUMMARY:
This study is a multicentre, randomized, open label on comparison of pancreatic beta cell recovery and preservation of Vildagliptin 100mg daily and Metformin (1000 - 2500mg) daily for 96 weeks in 203 patients with type 2 diabetes that will be conducted in four centers in Chennai. The primary outcome measures will be to compare the effects of Vildagliptin versus Metformin on Pancreatic beta cell function in type 2 diabetic patients as measure by Insulin secretion rate (ISR) relative to glucose0-2hr (pmol/min/m2/mmol/L). The secondary outcomes will be effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of Percent HbA1c reduction, C-peptide responses, Insulin to glucose ratios, Reduction in fasting plasma glucose (FPG), 2hr postprandial glucose (PPG) from baseline, Improvement in insulin sensitivity, Improvement in oral disposition index, Percentage of patients reaching the glycemic target of (i) HbA1c ≤ 6.5% and (ii)HbA1c ≤ 7.0%, in the overall study population and General safety in terms of occurrence of adverse events

DETAILED DESCRIPTION:
The subjects will be invited to the study center from the local population who are willing to participate in the trial. Each subject will be informed both orally and in writing about the study prior to inclusion in the study and only the subjects who give written informed consent will be included. The selection of the subjects is based on the inclusion and exclusion criteria defined in the protocol. The selected subjects will be given a screening number and subjected to screening procedure to find out eligible candidates for enrollment. The screening procedure includes obtaining subject's anthropometric data, baseline symptomatology, medical history, physical examination, laboratory investigations like blood glucose (fasting, 30min & 2hr after meal), HbA1c, ^Plasma insulin (fasting, 30min & 2hr after meal), ^2hr C peptide, Serum Amylase, Lipase, Urea, Creatinine, Gamma-glutamyl transferase (GGT), Urine albumin/creatinine ratio and urine pregnancy (if applicable).

The selected subjects after the screening procedure will be given a subject number and randomized between two arms. In Arm 1 they will be advised to take Vildagliptin 100mg daily for 96 weeks. In Arm 2 they are assigned Metformin (1000mg - 2500 mg/ day according to physician's preference for 96 weeks and all the subjects will be asked to come for follow up on week 12, week 24, week 48, week 72 and week 96. Subjects will be given sufficient quantity of study drugs. They will be instructed to take one tablet of Vildagliptin 50mg per day, 30 minutes after breakfast in the morning and second tablet at night, 30 minutes after dinner or Metformin tablets as per instructions given by the physician. Subjects will be instructed to maintain the record of dosing details in the patient diary.

Blood samples will be taken for the investigations such as blood glucose (fasting, 30min & 2hr after meal), HbA1c, Plasma insulin (fasting, 30min & 2hr after meal), C peptide (2hr after meal), fasting serum Amylase, Lipase, Urea, Creatinine, GGT, Urine albumin/creatinine ratio and Urine pregnancy test(if required) as specified in visit chart below. There will be three telephonic visits on week 36, week 60 and week 84. During those visits subject will be inquired about the health status over the phone and the drugs for the next three months will be dispensed by courier or delivered at home by the coordinator.

If the glycaemic control is constantly not satisfactory (HbA1c ≥ 8.5%) from visit 3, a rescue drug (Glimepiride) will be added to both arms and all the clinical and biochemical test will be done as per visit chart. With Glimepiride if the A1C is >9% insulin will be added and the subject will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Newly Diagnosed Type 2 Diabetes Mellitus patients not receiving any medication for diabetes
* HbA1c ranging from 7.0% to ≤ 8.5%
* Body Mass Index (BMI) ≥ 19.0 to ≤ 25.0 kg/m2
* Male and female subjects of age between 20 - 60 years shall be selected
* Adult subjects willing to give informed consent
* Subject must be available for and willing to attend all evaluation visits
* Willingness to follow the protocol requirements as evidenced by written informed consent
* Subject must have access to telephone for calling into the clinical center as part of test product compliance

Exclusion Criteria:

* Type 1 diabetes
* BMI ≤18.99 kg/m2 or> 25 kg/m2
* Presence of severe vascular complications
* Indications for use of insulin
* Elevated serum levels of lipase and amylase (>1.5 ULN)
* Gamma-glutamyltransferase >2 times upper limit of normal (ULN) at Visit1, confirmed by repeated measure within 3 working days
* Urine albumin: creatinine ratio (UACR) >1800 mg/g (>203.4 mg/mmol)
* Subjects below the age of 20 years and above the age of 60 years
* History of any drug abuse in the past 12 months
* History of hypersensitivity to study drugs and related drugs or excipients in the formulation.
* History of allergy to vegetables and or food substances and or any other manifestations suggestive of hypersensitivity reactions
* Subject who is not willing to participate in the study
* Clinically significant abnormal laboratory results at screening.
* Subject is being treated for severe active infection of any type
* A female subject who is breast-feeding, pregnant, or intends to become pregnant during the study
* Subject with clinically relevant uncontrolled medical condition (e.g hematologic renal hepatic neurology cardiac or respiratory)
* Subject has evidence of active malignancy, or prior history of active malignancy that has not been in remission for at least 5 years
* Participating in a clinical research trial within 30 days prior to screening
* Donated blood 3 months prior to first study visit and during the study period
* Individuals who are cognitively impaired and or who are unable to give informed consent
* Known HIV or Hepatitis B or C positive
* Any other health or mental condition that in the Investigator's opinion may adversely affect the subjects ability to complete the study or its measures or that may pose significant risk to the subject

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes in Insulin secretion rate | Baseline and 96 weeks
  To compare the effects of Vildagliptin versus Metformin on Pancreatic beta cell function in type 2 diabetic subjects as measure by Insulin secretion rate (ISR) relative to glucose0-2hr (pmol/min/m2/mmol/L)

SECONDARY OUTCOMES:
Changes in HbA1c reduction | Baseline and 96 weeks
  Effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of Percent HbA1c reduction
Changes in C peptide response | Baseline and 96 weeks
  Effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of C peptide response
Changes in Insulin to glucose ratio | Baseline and 96 weeks
  Effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of insulin to glucose ratio
Changes in Fasting plasma glucose | Baseline and 96 weeks
  Effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of reduction in fasting plasma glucose
Changes in 2hr postprandial plasma glucose | Baseline and 96 weeks
  Effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of reduction in 2hr postprandial plasma glucose
Changes in Insulin sensitivity | Baseline and 96 weeks
  Effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of improvement in insulin sensitivity
Changes in Oral disposition index | Baseline and 96 weeks
  Effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of improvement in oral disposition index
Percentage of subjects reaching HbA1c ≤ 6.5% | Baseline and 96 weeks
  Effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of percentage of subjects reaching the glycemic target of HbA1c ≤ 6.5%
Percentage of subjects reaching HbA1c ≤ 7.0% | Baseline and 96 weeks
  Effect of Vildagliptin versus Metformin based treatment on glycaemic variables in terms of percentage of subjects reaching the glycemic target of HbA1c ≤ 7.0%
Number of participant treated related to adverse event | Baseline and 96 weeks
  Number of adverse event observed in both Vildagliptin and Metformin treatment group will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ambady Ramachandran, MD,Ph.D,D.Sc, Principal Investigator — President, India Diabetes Research Foundation
Locations (6):
- India (6):
  - Jnana Sanjeevini Medical Centre, Bangalore, Karnataka
  - Vikas Pai Research Foundation, Pune, Maharashtra
  - Singhvi Health Centre, Chennai, Tamil Nadu
  - Dr V.Seshiah Diabetes research Institute, Dr V.Balaji Diabetes care centre, Chennai, Tamil Nadu
  - Arthur Asirvatham Hospital, Madurai, Tamil Nadu
  - Ramana Maharishi Rangammal Hospital, Tiruvannamalai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595